CLINICAL TRIAL: NCT05870280
Title: Nurse Coaching Given According to Integrative Nurse Coaching Theory the Effect of on Glisemic Control, Fear of Hypoglycemia and Risk Perception in Adults With Type 1 Diabetes.
Brief Title: Nurse Coaching the Effect of on Glycemic Control, Fear of Hypoglycemia and Risk Perception in Adults With Type 1 Diabetes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tuğba Bilgehan (Other)
Responsible Party: Sponsor-Investigator, Tuğba Bilgehan, Asst Prof, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TUGBABILGEHAN1
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Nurse's Role; Diabetes Mellitus; Hypoglycemia
Keywords: nurse coaching; diabetes; nursing
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RESPONSE GROUP (Experimental): After signing the voluntary consent form, the participants will be filled in the socio-demographic data collection form, the hypoglycemic attudes and behavior scale, the risk perception scale. A total of 4 group nurse coaching meetings will be held with individuals with type 1 diabetes, one to one over 7 days, under the framework of Theory of Integrative Nurse Coaching. Each of these interviews will last an average of 40-60 minutes. Interviews will be held online through the Zoom® webconferencing program at times scheduled jointly with the client. After the coaching meetings are over, the scales will be filled again and the HbA1c level will be requested from the blood results ordered at the doctor's request. In the coaching interviews, the materials specific to the coaching training received by the researchers (techniques such as the wheel of life, imagination, sabotage work, strong questions, Cartesian questions, SWOT analysis) will be used.
  Interventions: Behavioral: nurse coaching

INTERVENTIONS:
Behavioral: nurse coaching — Group coaching will be applied to individuals with diabetes, 5-8 people.

SUMMARY:
Because of the unforeseen rate of increase in case numbers, the high rates of mortality and morbidity, and the increased socio economic load it causes, diabetes has become the most discussed chronic and widespread metabolic disease in Turkey, and throughout the World, there are focused efforts to find a solution. It is very important for a person to self-assesss and evaluate to draw a roadmap for improved outcomes in a disease with a high financial and moral burden. A nurse is not only a caregiver to patients, but also a person who guides them to increased engagement and motivation in the care of their illness. Integrative Nurse Coaching is gaining notoriaty as an effective method to improve patient engagament and motivation in self-responsibility for health. The Integrative Nurse Coach Academy in the USA carries out studies and trainings to further this improvement. With cooperation between United States and Turkish nurse colleagues, it aims to bring Integrative Nurse Coach practice to Turkey. The Integrative Nurse Coach uses the nursing process as a framework to guide nurse coaching practice. This requires a shift in traditional nursing terminology and meaning to understand and incorporate the patient's subjective experience as follows: from assessment to stablishing a relationship, identifying readiness for change and the resources available to the patient for change; from nursing diagnosis to identifying opportunities and issues; from outcomes to having the patient set the agenda for achievement of the patient's goals; from 3 planning to creating the structure of the coaching interaction; from intervention to empowering the patient to reach goals; and from evaluating to assisting the patient to determine the extent to which goals were achieved.

The Theory of Integrative Nurse Coaching (TINC) , developed by the Integrative Nurse Coach Association , sheds light on this point. The TINC encompasses many holistic nursing theories and contains three concepts and five components. The three concepts are healing, metaparadigm in nursing theory (nurse, person, health, environment), and patterns of knowing in nursing (personal, empirics, aesthetics, ethical, not knowing, sociopolitical. The TINC five components include Integrative Nurse Coach Self-Development (self-reflection, self-assessment, self-evaluation self-care), Integral Perspective and Change, Integrative Lifestyle Health and Well-Being, Awareness and Choice, and Listening With Heart The five components all have equal value and form the basis for the nurse coach professional practice model. There is a parallel process of self-development for both the nurse coach and the client. The SelfDevelopment component empowers individuals (including the nurse coach) to focus on their health and wellness from an integral perspective and to identify their individual knowledge, expertise, strengths, and resources, while recognizing the fluidity of the change. The TINC is designed to guide nurse coaching practice, education, research, and health care policy. The theory emphasizes, describes, and directs the practice of nurse coaching, a recognized holistic nursing modality. It has been seen that the TINC framework is very suitable for individuals with diabetes to provide their own management.

DETAILED DESCRIPTION:
This research is a quasi-experimental study in pretest-posttest design research; It will be conducted with individuals with Type 1 diabetes who applied to Ankara City Hospital Endocrine Polyclinic. The sample size required for the study was found to be 95% power at 95% confidence level and 35 individuals for high-level effect size (f=0.40). However, the aim is to reach 40 individuals with the thought that data loss may occur during the study process.

Inclusion Criteria for Research; The patient;

* Being between the ages of 18-65,
* Having a smart phone and being able to use it actively,
* Having been diagnosed with type 1 diabetes at least 1 year ago,
* HbA1c > 7,
* Absence of any psychiatric or mental problems,
* Having the cognitive competence to answer the questions,
* Being able to speak, understand and read and write Turkish
* Patients who voluntarily agreed to participate in the study were included in the study.

Hypotesis H0: Nurse coaching given to individuals with Type 1 Diabetes has no effect on glycemic control, fear of hypoglycemia, and risk perception.

H1: Nurse coaching given to individuals with Type 1 Diabetes has an effect on glycemic control, fear of hypoglycemia and risk perception.

Data collection tools Data will be collected through the Sociodemographic data collection form, the hypoglycemıc attıtudes and behavıor scale, the risk perception scale.

Sociodemographic data collection form:

The form created by the researcher consists of questions about the sociodemographic information of the individual. In this section, besides questions about diabetes, there are questions such as gender, weight, height, age, marital status, educational status, occupation, economic status, and place of residence. The hypoglycemıc attıtudes and behavıor scale: The scale was developed by Polonsky. The 14-item 5-point Likert-type scale has 3 sub-dimensions. Anxiety, confidence, avoidance. The score of the sub-dimensions is calculated by dividing the number of items.

The risk perception scale: The scale was developed in 2007 and tested for validity and reliability. The scale is a self-report scale with 31 items that is easy to complete. Items 8,9,10,11,12, and 13 are scored inversely on the scale. The scale has 2 sub dimensions, namely risk knowledge and composite risk. These sub dimensions are evaluated separately in the scale and the total score from the scale is calculated through their total. The scores of the sub dimensions are calculated through dividing the total score by the number of items in the sub dimension.

ELIGIBILITY:
Inclusion Criteria:

The patient;

* Being between the ages of 18-65,
* Having a smart phone and being able to use it actively,
* Having been diagnosed with type 1 diabetes at least 1 year ago,
* HbA1c > 7,
* Absence of any psychiatric or mental problems,
* Having the cognitive competence to answer the questions,
* Being able to speak, understand and read and write Turkish
* Patients who voluntarily agreed to participate in the study were included in the study.

Exclusion Criteria:

* individual not participating in more than one interview
* unwillingness to quit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The hypoglycemıc attıtudes and behavıor | 1 month
  The 14-item 5-point Likert-type scale has 3 sub-dimensions. Anxiety, trust, avoidance. The score of the sub-dimensions is calculated by dividing the number of items.The highest score that can be obtained is 70 and the lowest score is 14.

SECONDARY OUTCOMES:
The risk perception | 1 month
  The scale is a self-report scale with 31 items that is easy to complete. Items 8,9,10,11,12, and 13 are scored inversely on the scale. The scale has 2 sub dimensions, namely risk knowledge and composite risk. These sub dimensions are evaluated separately in the scale and the total score from the scale is calculated through their total. The scores of the sub dimensions are calculated through dividing the total score by the number of items in the sub dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Bilgehan, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided